CLINICAL TRIAL: NCT05938010
Title: Subjective Wearing Experience of the Total30 for Astigmatism Lens Among Satisfied Biofinity Toric Lens Wearers
Status: Completed | Type: Observational
Sponsor: Scripps Poway Eyecare and Optometry (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: JM-23-01
Record Dates: First submitted 2023-06-30; First posted 2023-07-10 (Actual); Results first posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-08

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Dailies Total1® contact lenses for astigmatism (T30fA): Dailies Total1® contact lenses for astigmatism (T30fA)
  Interventions: Device: Dailies Total1® contact lenses for astigmatism (T30fA)

INTERVENTIONS:
Device: Dailies Total1® contact lenses for astigmatism (T30fA) — Dailies Total1® contact lenses for astigmatism (T30fA)

SUMMARY:
To subjectively evaluate wearing experience in the T30fA lens among subjects who were already satisfied with their Biofinity Toric lenses.

DETAILED DESCRIPTION:
This study is a single site, prospective, observational study of the subjective performance of T30fA in symptomatic patients. Subjects will be assessed at a screening visit, and 2 follow-up visits. Clinical evaluations will include measurement of visual acuity, manifest refraction, and patient questionnaires.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for the study if they meet the following criteria:

Note: Ocular criteria must be met in both eyes.

* Subjects who are currently wearing and can answer in the affirmative the following question: "I am satisfied with my current Biofinity toric monthly replacement lenses" prior to and after habitual lens optimization.
* Subjects between the ages of 18-45 who wear their Biofinity Toric lenses at least 5 days per week, at least 10 hours per day.
* Prescription with a sphere value between +4.00D and -6.00D inclusive, and a cylinder value between -0.75D and -2.25D.
* Vision Correctable to 20/20 (0.0 logMAR) or better in each eye at 6M with their Manifest refraction.
* Willing to attend all study visits.

Exclusion Criteria:

If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

* Ocular anterior segment infection, inflammation, abnormality, or active disease that would contraindicate contact lens wear.
* Use of systemic or ocular medications for which contact lens wear could be contraindicated as determined the investigator.
* Monocular (only 1 eye with functional vision) or fit with only 1 lens (and those patients that cannot be successfully fit with the T30fA lens design).
* Fitted with monovision.
* Prior ocular surgery.
* History of herpetic keratitis, ocular surgery, or irregular cornea.
* Pregnant or lactating.

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates they are unsuitable for the trial.

Pregnancy has a known effect on the stability of refractions and visual acuity. As such, subjects who become pregnant during the study will not be discontinued but their data may be excluded from analyses of effectiveness.

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Eligible participants will be 18-45 years of age who are current Biofinity Toric wearers and appropriate candidates for contact lens wear.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Mashouf, OD, Principal Investigator — Scripps Poway Eyecare & Optometry
Locations (1):
- Scripps Poway Eyecare & Optometry, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dailies Total1® Contact Lenses for Astigmatism (T30fA)
Started | 42
Completed | 40
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Dailies Total1® Contact Lenses for Astigmatism (T30fA)
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction With Comfort of T30fA Lens
Description: Subjects will give a rating between 0 and 10 (with 0 indicating not satisfactory at all and 10 indicating extremely satisfactory) best describing their comfort.
Time Frame: After 1 month of wear
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dailies Total1® Contact Lenses for Astigmatism (T30fA)
Number analyzed (Participants) | 40
score on a scale | 8 [7 to 9]

2. Other Pre Specified Outcome: Satisfaction With Visual Performance of T30fA Lens
Description: as for outcome 1
Time Frame: After 1 month of wear
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dailies Total1® Contact Lenses for Astigmatism (T30fA)
Number analyzed (Participants) | 40
score on a scale | 8 [8 to 9.3]

3. Other Pre Specified Outcome: Satisfaction With End of Day Comfort of T30fA Lens
Description: as for outcome 1
Time Frame: After 1 month of wear
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dailies Total1® Contact Lenses for Astigmatism (T30fA)
Number analyzed (Participants) | 40
score on a scale | 7 [4.7 to 8]

4. Other Pre Specified Outcome: Satisfaction With Ease of Handling of T30fA Lens
Description: as for outcome 1
Time Frame: After 1 month of wear
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dailies Total1® Contact Lenses for Astigmatism (T30fA)
Number analyzed (Participants) | 40
score on a scale | 9 [8 to 10]

5. Other Pre Specified Outcome: Satisfaction Overall of Handling of T30fA Lens
Description: as for outcome 1
Time Frame: After 1 month of wear
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dailies Total1® Contact Lenses for Astigmatism (T30fA)
Number analyzed (Participants) | 40
score on a scale | 8 [7 to 9]

ADVERSE EVENTS:
Time Frame: 4 weeks of lehfilcon A wear
Arm/Group | Dailies Total1® Contact Lenses for Astigmatism (T30fA)
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT05938010/Prot_SAP_000.pdf